CLINICAL TRIAL: NCT03618355
Title: Phase Ib Trial of Encapsulated Rapamycin (eRapa) in Prostate Cancer Patients Under Active Surveillance
Brief Title: Trial of eRapa in Prostate Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rapamycin Holdings, Inc. dba Emtora Biosciences (Industry)
Collaborators: Cancer Insight, LLC (Industry)
Responsible Party: Sponsor
Organization: Rapamycin Holdings Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RHI-P01
Record Dates: First submitted 2018-06-12; First posted 2018-08-07 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Oral administration with consecutive enrollment of overlapping dose-escalation cohorts, total treatment period 3 months. Patients will conclude treatment with previously scheduled standard of care prostate biopsy. With a single site screening patients into the cohorts at a rate of 3 patients every 6 weeks (4 weeks dosing and 2 weeks safety assessment), a new cohort will start approximately every 6 weeks. Therefore, if each cohort of 3 patients are pre-screened and there are no dose limiting toxicities (DLT), the 4th and final dose cohort will be enrolled at approximately 18 weeks. Each patient will be on study for 6 months; therefore, 10-11 months will be the shortest time for trial completion. Given unforeseen delays, we anticipate the trial to take approximately one year to complete.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: 0.5 mg weekly (Experimental): Oral administration with consecutive enrollment of overlapping dose-escalation cohorts, total treatment period 3 months. Patients will conclude treatment with previously scheduled standard of care prostate biopsy.
  eRapa (encapsulated rapamycin) is dosed at 0.5 mg every week.
  Interventions: Drug: eRapa (encapsulated rapamycin)
- Cohort 2: 1 mg weekly (Experimental): Oral administration with consecutive enrollment of overlapping dose-escalation cohorts, total treatment period 3 months. Patients will conclude treatment with previously scheduled standard of care prostate biopsy.
  eRapa (encapsulated rapamycin) is dosed at 1 mg every week.
  Interventions: Drug: eRapa (encapsulated rapamycin)
- Cohort 3: 0.5 mg daily (Experimental): Oral administration with consecutive enrollment of overlapping dose-escalation cohorts, total treatment period 3 months. Patients will conclude treatment with previously scheduled standard of care prostate biopsy.
  eRapa (encapsulated rapamycin) is dosed at 0.5 mg daily.
  Interventions: Drug: eRapa (encapsulated rapamycin)
- Cohort 4: 1 mg daily (Experimental): Oral administration with consecutive enrollment of overlapping dose-escalation cohorts, total treatment period 3 months. Patients will conclude treatment with previously scheduled standard of care prostate biopsy.
  eRapa (encapsulated rapamycin) is dosed at 1 mg daily.
  Interventions: Drug: eRapa (encapsulated rapamycin)

INTERVENTIONS:
Drug: eRapa (encapsulated rapamycin) — The eRapa (encapsulated rapamycin) drug product consists of sub-micron rapamycin particles incorporated into poly(methyl methacrylate) polymer (Eudragit® L 100 / S 100).
  This improved formulation and better bioavailability enables eRapa to consistently provide approximately 30% more drug than sirolimus (unpublished data). Improved and predictable delivery allows for consistent and sustained lower dosing, which will result in an improved toxicity profile since the latter is proven to be related to blood concentration levels. This is a phase Ib trial in low risk (Gleason score ≤7 (3+4)) prostate cancer patients under active surveillance to establish dosage safety and treatment levels.

SUMMARY:
This study is to determine the safety, pharmacokinetics/pharmacodynamics, and immunologic impact of encapsulated rapamycin in patients with low risk prostate cancer under active surveillance. There will be four groups of patients, each receiving a different dose of rapamycin.

DETAILED DESCRIPTION:
This is a phase Ib trial of encapsulated rapamycin to determine safety, pharmacokinetics/pharmacodynamics, and immunologic impact in patients with low risk prostate cancer under active surveillance. This new formulation, encapsulated rapamycin (sirolimus), provides a more predictable bioavailability of this drug than [the other formulation]. The encapsulated and targeted rapamycin (eRapa) can be delivered at a consistent and lower dosage, not only improving the toxicity profile but also capitalizing on the newly appreciated mechanism of partial and/or intermittent mTOR inhibition, making eRapa an ideal immuno-oncologic and chemopreventative agent. Low dose rapamycin has been shown to prevent cancer formation, progression, and/or recurrence in the majority of cancer histologies including the most prevalent: lung, breast, prostate, and colon cancers.

ELIGIBILITY:
Inclusion Criteria:

-

The patient must:

* Have pathologically (histologically) proven diagnosis of prostate cancer with a Gleason score ≤7 (3+4) and already undergoing active surveillance
* Be able to give informed consent
* Be age 18 or older

Exclusion Criteria:

* Prostate cancer with a Gleason score >7
* Unable to give informed consent
* Age < 18
* Immunosuppressed state (e.g., HIV, use of chronic steroids)
* Active, uncontrolled infections
* On medications with strong inhibitors or inducers of CYP3A4 and or P-gp.
* On agents known to alter rapamycin metabolism significantly (Appendix H)
* Have another cancer requiring active treatment (except basal cell carcinoma or squamous cell carcinoma of the skin)
* Individuals with a reported history of liver disease (e.g., cirrhosis)
* Individuals who are not a good candidate for active surveillance in their treating physician's opinion
* Have a medical condition (e.g., anemia, anticoagulated) for which repeated phlebotomy may be problematic.
* Uncontrolled hypertension.
* Individuals that have abnormal screening vital organ function prior to enrollment

  * Liver Function Test

    * Bilirubin >2.0
    * Alkaline phosphatase >5x upper limit of normal (ULN)
    * ALT/AST >2x ULN
  * Complete Blood Count:

    * WBC elevated above the normal standard per the testing laboratory
    * Hgb/Hct below the normal standards of the testing lab
    * Platelets below the normal standards of the testing lab
  * Total Cholesterol >240 mg/dL
  * Triglycerides > 200 mg/dL
  * Serum creatinine >2 and BUN >30
  * Urinary protein: proteinuria >1+ on urinalysis or >1 gm/24hr

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patient must have pathologically (histologically) proven diagnosis of prostate cancer with a Gleason score ≤7 (3+4) and already undergoing active surveillance.
Enrollment: 15 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2019-12-02 (Actual)

PRIMARY OUTCOMES:
Primary Safety and Tolerability (Incidence of Treatment-Emergent Adverse Events) | After 4 weeks of treatment in each dosing cohort.
  To analyze the overall safety of eRapa by evaluating the number, frequency, duration, and relation of toxicity events as defined by the Common Terminology Criteria for Adverse Events (CTCAE) v4.03.
Primary Safety and Tolerability (Incidence of Treatment-Emergent Adverse Events) | After completion of treatment, approximately 12 weeks, in each dosing cohort.
  To analyze the overall safety of eRapa by evaluating the number, frequency, duration, and relation of toxicity events as defined by the Common Terminology Criteria for Adverse Events (CTCAE) v4.03.
Primary Safety and Tolerability (Incidence of Treatment-Emergent Adverse Events) | This will be completed after all dosing cohorts have been enrolled and treated, anticipated to occur at 1 year.
  To compare safety between dosing cohorts of eRapa by evaluating the number, frequency, duration, and relation of toxicity events as defined by the Common Terminology Criteria for Adverse Events (CTCAE) v4.03 at the 4 week time point.
Primary Safety and Tolerability (Incidence of Treatment-Emergent Adverse Events) | This will be completed after all dosing cohorts have been enrolled and treated, anticipated to occur after 1 year.
  To compare safety between dosing cohorts of eRapa by evaluating the number, frequency, duration, and relation of toxicity events as defined by the Common Terminology Criteria for Adverse Events (CTCAE) v4.03 at the 12 week time point.

SECONDARY OUTCOMES:
Secondary Pharmacokinetics: AUC | Cohorts 1 and 2 PK analysis will occur during the first week. Cohorts 3 and 4 PK analysis will occur during week 12 of treatment.
  Pharmacokinetics of eRapa in blood will be evaluated throughout the trial and compared within and between the dosing cohorts. For cohorts 1 and 2, single dose exposure curves will be generated by assessing the rapamycin levels in whole blood and spot card collection at 0, 0.5, 1, 2, 4, 6, 8, 24, 48, and 72 hrs after the first dose on week 1. Cohorts 3 and 4, exposure curves will be generated during the last week of treatment with blood draws and spot card collection after a dose during the final week at 0, 0.5, 1, 1.5, and 2 hrs.
Secondary Pharmacokinetics: Exposure Trough Levels | Cohorts 3 and 4 PK analysis will occur during the first week of treatment.
  Pharmacokinetics of eRapa in blood will be evaluated throughout the trial and compared within and between the dosing cohorts. Cohorts 3 and 4, eRapa troughs will be gathered before the first 5 doses of eRapa during the week 1.
Secondary Pharmacodynamics: mTOR inhibition in PBMC by assessment of phosphorylation of S6 | Cohorts 1 and 2 PD analysis will occur during the first week. Cohorts 3 and 4 PD analysis will occur during week 12 of treatment.
  Pharmacodynamics of eRapa in blood will be evaluated throughout the trial and compared within and between dosing cohorts. For cohorts 1 and 2, mTOR inhibition in PBMC by assessment of phosphorylation of S6 will also be assessed at 0, 0.5, 1, 2, 4, 6, 8, 24, 48, and 72 hrs after the first dose on week 1. Cohorts 3 and 4, mTor inhibitions will be gathered before the first 5 doses of eRapa during the week 1. In addition, during the last week of treatment after a dose during the final week at 0, 0.5, 1, 1.5, and 2 hrs.
Secondary Pharmacodynamics: mTOR inhibition upon initial dose | Cohorts 1 and 2 PD analysis will occur during the first week.
  Pharmacodynamics of eRapa in blood will be evaluated throughout the trial and compared within and between dosing cohorts. For cohorts 1 and 2, mTOR inhibition in PBMC by assessment of phosphorylation of S6 will also be assessed at 0, 0.5, 1, 2, 4, 6, 8, 24, 48, and 72 hrs after the first dose on week 1.
Secondary Pharmacodynamics: mTOR inhibition first week of daily dosing | Cohorts 3 and 4 PD analysis will occur during week 12 of treatment.
  Pharmacodynamics of eRapa in blood will be evaluated throughout the trial and compared within and between dosing cohorts. For cohorts 3 and 4, mTOR inhibition in PBMC by assessment of phosphorylation of S6 will also be assessed before the first 5 doses of eRapa during the week 1.
Secondary Pharmacodynamics: mTOR inhibition during final week of treatment | Cohorts 3 and 4 PD analysis will occur during week 12 of treatment.
  Pharmacodynamics of eRapa in blood will be evaluated throughout the trial and compared within and between dosing cohorts. For cohorts 3 and 4, mTOR inhibition in PBMC by assessment of phosphorylation of S6 will also be assessed during the last week of treatment after a dose during the final week at 0, 0.5, 1, 1.5, and 2 hrs.
Secondary Immunologic Response: T cell phenotype individually | Assessments will occur at baseline, during (after 4 weeks), after short-term completion of treatment (after 12 weeks), and long-term completion of treatment (6 months).
  Immunologic response will be measured and compared from baseline at specified time points throughout the trial. The specific analysis of T cell naïve/memory/effector phenotype. These results will be assessed individually.
Secondary Immunologic Response: T cell function individually | Assessments will occur at baseline, during (after 4 weeks), after short-term completion of treatment (after 12 weeks), and long-term completion of treatment (6 months).
  Immunologic response will be measured and compared from baseline at specified time points throughout the trial. The specific analysis of T cell exhaustion markers (PD-1, LAG3, TIM3), and homing markers (CD62L, CCR7). These results will be assessed individually.
Secondary Immunologic Response: T cell phenotype within each dosing cohort | Assessments will occur at baseline, during (after 4 weeks), after short-term completion of treatment (after 12 weeks), and long-term completion of treatment (6 months).
  Immunologic response will be measured and compared from baseline at specified time points throughout the trial. The specific analysis of T cell naïve/memory/effector phenotype. These results will be assessed within each dosing cohort.
Secondary Immunologic Response: T cell function within each dosing cohort | Assessments will occur at baseline, during (after 4 weeks), after short-term completion of treatment (after 12 weeks), and long-term completion of treatment (6 months).
  Immunologic response will be measured and compared from baseline at specified time points throughout the trial. The specific analysis of T cell exhaustion markers (PD-1, LAG3, TIM3), and homing markers (CD62L, CCR7). These results will be assessed within each dosing cohort.
Secondary Immunologic Response: T cell phenotype overall study-wide | Assessments will occur at baseline, during (after 4 weeks), after short-term completion of treatment (after 12 weeks), and long-term completion of treatment (6 months).
  Immunologic response will be measured and compared from baseline at specified time points throughout the trial. The specific analysis of T cell naïve/memory/effector phenotype. These results will be assessed overall study-wide.
Secondary Immunologic Response: T cell function overall study-wide | Assessments will occur at baseline, during (after 4 weeks), after short-term completion of treatment (after 12 weeks), and long-term completion of treatment (6 months).
  Immunologic response will be measured and compared from baseline at specified time points throughout the trial. The specific analysis of T cell exhaustion markers (PD-1, LAG3, TIM3), and homing markers (CD62L, CCR7). These results will be assessed overall study-wide.
Secondary Quality of Life Analysis | Assessments performed baseline, after completion of therapy (approximately 12 weeks), and after 6 months.
  Quality of life will be assessed and compared to characterize the impact of eRapa before, during, and after treatment by using the National Institute of Health Patient-Reported Outcomes Measurement Information System (PROMIS-29) and Cognition (long form) assessments.

CONTACTS AND LOCATIONS:
Overall Officials: George E Peoples, MD, FACS, Study Director — Cancer Insight
Locations (1):
- UT Health San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No